CLINICAL TRIAL: NCT00262613
Title: Long-Term Use of Inhaled Sodium Pyruvate for the Treatment of Chronic Obstructive Pulmonary Disease
Brief Title: Sodium Pyruvate Therapy in COPD Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emphycorp (Industry)
Collaborators: Cellular Sciences, inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSI-NII5-021
Record Dates: First submitted 2005-12-06; First posted 2005-12-07 (Estimated); Last update posted 2006-05-29 (Estimated); Status verified 2006-05

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Sodium Pyruvate; COPD; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Sodium Chloride

INTERVENTIONS:
Drug: sodium pyruvate in 0.9% sodium chloride solution

SUMMARY:
In animal models, sodium pyruvate has been shown to be an effective anti-inflammatory agent, and in human studies sodium pyruvate has been shown to be a bronchodilating agent. Subjects with COPD are known to have inflammation in the lung, and often have bronchoconstriction. As such, these subjects typically are on multiple therapies, including steroid therapy. This trial will study the effect of inhaled sodium pyruvate on inflammation and lung function in COPD subjects over a six week period.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a disease, which involves the conducting airways of the respiratory tract and affects 5-10% of individuals in the United States. The morbidity and mortality associated with this disease are increasing both in the United States and worldwide (1). The mechanisms involved in the pathogenesis of COPD are complex but it can be classified as an inflammatory disease of the airways characterized by an increase in inflammatory cells (neutrophils, macrophages, and lymphocytes) both in the bronchial mucosa and in bronchoalvaeolar lavage fluid (2). Some of the many therapeutic approaches to managing this disease include various inhaled compounds, such as, bronchodilators (i.e. beta agonists) and both inhaled and systemic steroid treatment. The current therapies are not without adverse side effects. The purpose of this study is to test the safety and therapeutic value of an endogenous compound, sodium pyruvate, with anti-inflammatory properties (anti-oxidant) in patients with COPD.

Reactive oxygen species (ROS), such as superoxide anion, free hydroxyl radical, and hydrogen peroxide, have been shown to be toxic to various mammalian tissue (3), including lung (4--6), and have been implicated in many human diseases (7). Anti- oxidant therapy has been shown to be effective in several animal models of inflammatory lung diseases (8-10). Sodium pyruvate is a part of the body's natural endogenous anti-oxidant defense system. It is secreted by cells, readily enters cells, and can react with peroxide to "detoxify it (11-13). Since hydrogen peroxide is also a precursor to other ROS, inhibition of it has broad anti-oxidant effects. Sodium pyruvate has been shown to have protective anti-oxidant activity both in vitro (11, 14-17) and in vivo (18, 19).

Clinically, sodium pyruvate has been given to patients for a variety of disorders ranging from Friedreich's ataxia (20) to open heart operations (21). It has been administered via several routes including intravenous (20-23), topical administration for hyperkeratotic disorders (24), and in dietary supplementation (25-29). Animal model studies in rats and rabbits were conducted to assess potential adverse effects. Rats were used to assess the impact of sodium pyruvate administered directly to the lungs by intratracheal injection (Rat Study). Rabbits were used to assess the impact of sodium pyruvate administered as an inhaled mist using a nebulizer (Pyruvate Inhalation Study in Rabbits). There were no adverse effects noted in the parameters, which were monitored for acute lung injury (histology, bronchoalveolar lavage fluid content, and arterial blood gas analysis). In addition, it was shown that the intratrachcheal administration of sodium pyruvate was beneficial in diminishing the development of acute lung injury in rats induced by bleomycin. The generation of toxic oxygen radicals is believed to be a major mechanism of bleomycin lung toxicity.

There are two major groups of COPD medications: 1) Bronchodilator agents that inhibit the bronchoconstriction characteristic of some patients with COPD; and 2) anti-inflammatory agents which inhibit the inflammatory components responsible for the airway narrowing and increased mucus production, also characteristic features of patients with COPD. The known anti-oxidant properties of sodium pyruvate make it an attractive compound for possible therapeutic efficacy, which should have in vivo anti-inflammatory effects. In addition to its possible anti-inflammatory properties, we previously observed (Phase I study of this compound, see Phase I report) acute therapeutic efficacy in patients with mild bronchial asthma. The observed improvement in FEV1 at 30 minutes to 2 hours post inhalation of sodium pyruvate suggests a bronchodilator effect in these patients. The mechanism of action is unclear at this time but it may be a result of the ability of inhaled sodium pyruvate to modulate reactive oxygen and nitrogen species such as H2O2 and nitric oxide (NO). These species have both been shown to be elevated in expired breath of patients with COPD and asthma and thus implicated in the pathogenesis (30-39). Nitric oxide has been shown to play an important role in maintaining normal physiologic homeostasis in the normal and injured lung (40-42). It has been shown to reverse acetylcholine and histamine induced bronchoconstriction and to maintain normal vascular integrity (40-42). It is possible that inhaled sodium pyruvate alters airway levels of both oxygen and nitrogen reactive species resulting in a beneficial effect.

Since sodium pyruvate is endogenous, has been used previously in patients, had no adverse affects in our animal model studies, and had no adverse effects in our acute Phase I Clinical Trial in patients with mild bronchial asthma, we feel that we will be able to use it safely in this long term multiple use study in patients with COPD. For safety considerations only the lowest concentration of sodium pyruvate (0.5mM) studied previously in our single dose Safety Trial will be studied in this 3-times/day double blind placebo controlled 6 week study. The total daily dose per subject will be similar to the 1.5mM concentration (3 doses of 0.5mM). In addition, it is approximately 3 times less than the total daily dose given to subjects who received the 5.0mM concentration in our Single Dose Phase I Safety Trial. The proposed study is designed to address both the long term multiple dose safety aspects of inhaled sodium pyruvate as well as both the acute and long-term efficacy of the compound. The acute study is designed to evaluate the possible bronchodilator effects and the long term multiple use study is designed to evaluate the anti-inflammatory properties of sodium pyruvate.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a clinical diagnosis of moderate to severe COPD, <70% predicted FEV1, and a stable pulmonary disease status.

Exclusion Criteria:

* a. Pulmonary disease other than COPD
* b. Clinically significant cardiac disease including uncontrolled congestive heart failure and unstable angina
* c. Pregnancy
* d. Females of child bearing potential age not on adequate contraception or lactating
* e. Subjects receiving oral or IV corticosteroid treatment within one month of Screening Visit
* f. Less than 18 years of age and greater than 85 years of age
* g. Hospitalization within last 6 months due to acute exacerbation of air-way disease
* h. Subjects on escalating dose of immunotherapy
* i. Subjects with a clinically significant abnormal chest x-ray within past 12 months.
* j. Medication changes within 1 month
* k. Subjects who have participated in another investigation drug treatment study within the previous month.
* l. Subjects with a current history of alcohol abuse or recreational drug use.
* m. Subjects who have taken vitamins with anti-oxidant properties (E or C) or dietary supplements containing pyruvate within 24 hours prior to the screening visit.
* n. Subjects who use less than 4 puffs of Albuterol a day over the period between the Screening Visit and Visit 1.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2004-09; Study Completion 2006-05

PRIMARY OUTCOMES:
Lung function, as determined by spirometry
Safety, as determined by laboratory analyses

SECONDARY OUTCOMES:
Levels of Nitric Oxide in expired air
Results of Chronic Respiratory Disease Questionnaire
SaO2 levels

CONTACTS AND LOCATIONS:
Overall Officials: John J. Votto, D.O., Principal Investigator — Hospital for Special Care
Locations (2):
- United States (2):
  - Hospital for Special Care, New Britain, Connecticut
  - Yale University School of Medicine, New Haven, Connecticut

REFERENCES:
- See also: Emphycorp Website — http://emphycorp.com